CLINICAL TRIAL: NCT06201117
Title: The Effects of Preparatory Information Using Digital Media on Anxiety and Treatment Adherence Behavior in Patients Undergoing Cardiac Surgery
Brief Title: Effects of Preparatory Information on Anxiety and Treatment Adherence in Heart Surgery Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Keattiwan Kansaard, Faculty of Nursing, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: HE661478
Record Dates: First submitted 2023-12-31; First posted 2024-01-11 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Heart Surgery
Keywords: Heart Surgery, Digital Media, Preparatory Information

STUDY DESIGN:
Intervention Model Description: 2-arm parallel randomized controlled trial study
Who Masked: Outcomes Assessor
Masking Description: The research assistants who are blinded for the participant groups evaluate the outcomes including anxiety, 30 minutes after the intervention or usual care and 48 hours after the surgery and treatment adherence 1 time, 48 hours after the surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preparatory information (Experimental): In the experimental group, the participants will rate their anxiety before receiving the 12-minute preparation information video in addition to the usual preparation information on the day they gave consent to participate in the study. The participants will rate their anxiety again 30 minutes after the intervention. The experimental group will receive the preparation video again the second time on the day before surgery. Anxiety and treatment adherence will be measured in the ICU, 48 hours after the surgery.
  Interventions: Behavioral: Preparatory information for ICU stay; Behavioral: Usual information
- Usual information (Active Comparator): In the comparison group, the participants will rate their anxiety before receiving the usual preoperative information on the day they gave consent to participate in the study. The participants will rate their anxiety again 30 minutes after the usual information. Anxiety and treatment adherence will be measured in the ICU, 48 hours after the surgery.
  Interventions: Behavioral: Usual information

INTERVENTIONS:
Behavioral: Preparatory information for ICU stay — Preparatory information for ICU stay after cardiac surgery via 12-minute digital media
  Arms: Preparatory information
Behavioral: Usual information — Preoperative information that is given to patients before having cardiac surgery

SUMMARY:
The goal of this clinical trial is to investigate the effects of providing information to prepare for ICU stay in patients after heart surgery on anxiety and cooperative behaviors. The main questions it aims to answer are:

* Are the anxiety levels before and after receiving prepared information video (VDO) and usual information different among participants in the experimental group?
* Are the anxiety levels between participants who received prepared information VDO and usual information and usual information only different?
* Are the cooperative behaviors during a recovery period in the ICU between participants who received prepared information VDO and usual information and usual information only different?

The researcher will provide the prepared information for ICU stay through 12-minutes VDO, 2 times before the surgery to the experimental group in addition to the usual pre-operative information (usual care). Participants in the comparison group will receive usual pre-operative information only to see if the anxiety and cooperative behaviors during a recovery period in the ICU differ between the groups.

DETAILED DESCRIPTION:
• Participant invitation The study invitation for the prospective participants who are patients scheduled for heart surgery is posted at the cardiothoracic surgery outpatient clinic. Before deciding, patients who are interested in participating can get in touch with the researchers to learn more about the study.

Additionally, the invitation will also be posted at the in-patient facilities where patients are being admitted for heart surgery so the nurses to ask patients for their interest in being the study volunteers. The researchers will be notified if there are potential participants.

* Recruitment and consent process The researcher will meet with prospective participants in in-patient units where they are being admitted for surgery to discuss the study details and evaluate the Abbreviated Mental Test for screening. Potential participants who have an AMT test score of less than 8 will be excluded and thanked for their volunteer. The consent will be signed by the patients who agree to participate. The meeting will take place between 6:00 and 8:00 p.m. after patients have completed all preoperative preparations and have had dinner.
* Research assistants Two research assistants in this study are registered nurses with more than 3 years of experience in caring for heart surgery patients. They were trained to follow the study protocol and use research instruments. The interrater reliability between the researchers and research assistants is 0.96. To avoid bias, the research assistants will evaluate the outcomes in both the experimental and comparison groups while remaining blind to group allocation.
* Sample size estimation The sample size estimation was calculated using the G*Power 3.1.9.7 program for a two-sample t-test for independent with 0.8 effect size from Cohen's d formula (Cohen, 1988) using mean anxiety from a similar study. The estimated sample size needed for this study is 21 for each group with 10% adjusted for attrition resulting in 24 participants necessary for each group to demonstrate an effect.
* Data collection Data collection starts once the participants sign the consent. The participants will be allocated to a group with computer computer-generated program. Allocation to the group cannot be concealed from the participants but will be blinded to the research assistants who evaluate the outcomes. In the experimental group, the researcher asks participants to rate their anxiety before receiving the intervention (12-minute preparation information video + usual preparation information) while in the comparison group, only usual preparation information is given. The participants rated their anxiety again 30 minutes after the intervention and the usual information was given. The experimental group will receive the preparation VDO again the day before surgery. Participants in both groups rate their anxiety 48 hours after surgery and are evaluated for treatment adherence during their ICU stay. Participants who are unable to participate until the completion of the trial for any reason will be withdrawn from the study and analysis. Individual participant identities will not be recorded or disclosed in any way. Data analysis will be used to identify groups, and all recorded information will be deleted two years after the study is completed.
* Data analysis The data analysis will be performed using the Statistical Package for the Social Sciences (SPSS) version 28 software with a confidence interval of 95% (α=0.05). Descriptive statistics, Chi-square test, ANOVA, and Mann-Whitney U test will be analyzed to evaluate demographic differences between the groups depending on the normality assumption. Repeated measures ANOVA and ANCOVA will be used to analyze differences in anxiety and treatment adherence within the groups and between the groups, respectively. However, if the normality assumption is not fulfilled, the Mann-Whitney U test and Chi-square will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Attending heart surgery as scheduled for the first time
2. Never been admitted to the intensive care unit.
3. Stable condition before surgery
4. Ability to understand communication in Thai
5. Willingness to participate in the study.

Exclusion Criteria:

1. Impaired cognitive ability: assessed by the Abbreviated Mental Test (AMT) when the score is less than 8 out of 10.
2. Admitted to the hospital in an emergency and need urgent surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-12-27 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Anxiety | Anxiety will be measured 3 times in both groups immediately before receiving preparatory information or usual information, 30 minutes after receiving preparatory information or usual information, and 48 hours after the surgery.
  The 1-Item Anxiety Visual Analogue Scale (AVAS) horizontal version is used to assess participants' level of perceived anxiety. AVAS is a numerical scale that is rated on a 10-centimeter linear scale, with 0 indicating no anxiety on the left end and 10 reflecting the most intense anxiety, representing a score of 100 on the right end.
Treatment adherence | The research assistants who are blinded for the participant groups evaluate the treatment adherence 1 time at 48 hours after the surgery.
  Treatment adherence is measured using the observational checklist developed by the researchers based on the content instructed in the preparatory information VDO. The checklist consists of 19 items in 4 categories including procedural adherence, sensory adherence, behavioral adherence, and coping adherence The checklist was evaluated by 5 experts and yielded a scale content validity index (S-CVI) of 1.0. The score of each item is rated as 0-2 scale where 0 means no adherence, 1 is partial adherence, and 2 is absolute adherence. The total possible score ranges from 0-57.

CONTACTS AND LOCATIONS:
Overall Officials: Dr.RACHATA MALA, 3, Study Chair — Faculty of medicine, KKU
Locations (1):
- Srinagarind Hospital, Khon Kean University, Khon Kaen, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Aardoom JJ, Loheide-Niesmann L, Ossebaard HC, Riper H. Effectiveness of eHealth Interventions in Improving Treatment Adherence for Adults With Obstructive Sleep Apnea: Meta-Analytic Review. J Med Internet Res. 2020 Feb 18;22(2):e16972. doi: 10.2196/16972. PMID 32130137
- [Result] Aust H, Eberhart L, Sturm T, Schuster M, Nestoriuc Y, Brehm F, Rusch D. A cross-sectional study on preoperative anxiety in adults. J Psychosom Res. 2018 Aug;111:133-139. doi: 10.1016/j.jpsychores.2018.05.012. Epub 2018 May 22. PMID 29935747
- [Result] Bowyer A, Jakobsson J, Ljungqvist O, Royse C. A review of the scope and measurement of postoperative quality of recovery. Anaesthesia. 2014 Nov;69(11):1266-78. doi: 10.1111/anae.12730. Epub 2014 Jun 2. PMID 24888412
- [Result] Cardiovascular thoracic intensive care unit. (2020). Srinagarind hospital adult cardiac surgery database: 2020 update.
- [Result] Dale JG, Midthus E, Dale B. Using information and communication technology in the recovery after a coronary artery bypass graft surgery: patients' attitudes. J Multidiscip Healthc. 2018 Aug 30;11:417-423. doi: 10.2147/JMDH.S175195. eCollection 2018. PMID 30214223
- [Result] Elgazzar SE, Qalawa SAA, Ali Hassan AM. Impact of educational programme on patient's health outcomes following open heart surgeries. Nurs Open. 2023 May;10(5):3028-3041. doi: 10.1002/nop2.1549. Epub 2022 Dec 8. PMID 36480022